CLINICAL TRIAL: NCT07037589
Title: Women With isoLated acUte cyStitis and Macroscopic Hematuria. Is Further Investigation Needed? A Prospective Multicenter Study. BLUSH Trial
Brief Title: Women With isoLated acUte cyStitis and Macroscopic Hematuria. Is Further Investigation Needed?
Acronym: BLUSH
Status: Recruiting | Type: Observational
Sponsor: Vastra Gotaland Region (Other Government)
Responsible Party: Sponsor
Other Study IDs: BLUSH trial
Record Dates: First submitted 2025-06-16; First posted 2025-06-25 (Actual); Last update posted 2025-11-21 (Actual); Status verified 2025-06

CONDITIONS: Hematuria; Acute Cystitis With Hematuria; Bladder Cancer; Urothelial Carcinoma; Renal Cancer
MeSH Terms: conditions — Hematuria; Urinary Bladder Neoplasms; Carcinoma, Transitional Cell; Kidney Neoplasms | interventions — Cystoscopy; Cytological Techniques

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- AHG (Acute Hemorrhagic Cystitis Group):: Patients with acute onset macroscopic hematuria with lower urinary tract symptoms such as dysuria, frequency, and urgency of less than one week's duration.
  Interventions: Procedure: investigation setting (cystoscopy + CTU + cytology)
- non AHG (non-Acute Hemorrhagic Cystitis Group):: Patients with atypical clinical presentation such as:
  Chronic irritative symptoms >4 weeks. Recurrent UTI (≥2 episodes in 6 months or ≥3 episodes per year). Febrile UTI. Absence of irritative symptoms.
  Interventions: Procedure: Cystoscopy - CTU - cytology (if needed)

INTERVENTIONS:
Procedure: investigation setting (cystoscopy + CTU + cytology) — Observational study. All patients in this group undergo standard diagnostic evaluation including cystoscopy, CT urography, and urine cytology (if clinically indicated), performed during initial assessment for acute macroscopic hematuria.
  Groups: AHG (Acute Hemorrhagic Cystitis Group):
Procedure: Cystoscopy - CTU - cytology (if needed) — All patients in this group undergo standard diagnostic evaluation including cystoscopy, CT urography, and urine cytology (if clinically indicated), performed during initial assessment for atypical or chronic presentations of macroscopic hematuria.
  Groups: non AHG (non-Acute Hemorrhagic Cystitis Group):

SUMMARY:
This prospective multicenter observational study evaluates whether women ≥50 years with isolated acute hemorrhagic cystitis (AHC) and macroscopic hematuria require full malignancy workup. All participants undergo standard diagnostics (cystoscopy, CT urography, cytology), with 12-month follow-up for cancer detection. The aim is to identify low-risk patients where invasive investigations may be safely avoided.

DETAILED DESCRIPTION:
The BLUSH trial is a prospective, multicenter, observational study investigating whether full malignancy workup is necessary in women ≥50 years presenting with isolated acute hemorrhagic cystitis (AHC) and macroscopic hematuria. AHC is defined as macroscopic hematuria accompanied by acute lower urinary tract symptoms (dysuria, frequency, urgency) of less than one week's duration. Women with prior urological malignancies, significant comorbidities, or impaired consent capacity are excluded.

All enrolled patients undergo standardized initial assessment including full clinical history (smoking, family history, comorbidities), physical examination, urinalysis, urine culture, cystoscopy, CT urography, and cytology when indicated. Participants are stratified into AHC and non-AHC groups based on symptomatology and laboratory findings. Data collection includes demographics, symptom duration, urine findings, cancer diagnoses (type, stage, grade), treatment details, and clinical outcomes.

Patients are followed for a minimum of 12 months via medical record review to capture delayed cancer diagnoses. Data are pseudonymized and stored securely under GDPR regulations. The primary outcome is the incidence of urological malignancy within one year. Secondary outcomes include time to diagnosis, proportion of avoidable invasive procedures, and accuracy of the AHC classification in predicting cancer risk.

The study aims to support individualized risk-based management in women with hematuria.

ELIGIBILITY:
Inclusion Criteria:

1. Women ≥50 years of age.
2. Macroscopic hematuria.
3. Presenting for evaluation within the SCP for macroscopic hematuria.
4. Ability to provide informed consent.

Exclusion Criteria:

1. Prior diagnosis of bladder cancer, renal cancer, or upper tract urothelial carcinoma (UTUC).
2. Cognitive impairment preventing informed consent.
3. Ongoing or recent treatment for urological malignancy.
4. Serious comorbidities affecting participation or safety.
5. Pregnant women.

Ages: 18 Years to 110 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Eligibility is limited to individuals identifying as female, based on self-reported gender identity.
Study Population: Women aged 50 years and older presenting with macroscopic hematuria. Participants are recruited at initial presentation within the standard care pathway for hematuria evaluation at participating centers in Sweden.
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2025-10-13 (Actual); Primary Completion 2026-08-30 (Estimated); Study Completion 2027-08-30 (Estimated)

PRIMARY OUTCOMES:
Incidence of urological malignancy | At least 12 months from study inclusion.
  The proportion of women diagnosed with urological cancer (bladder, upper urinary tract, or kidney cancer) within 12 months after initial presentation of macroscopic hematuria.

SECONDARY OUTCOMES:
Time to cancer diagnosis | At least 12 months from study inclusion.
  Duration from initial presentation to confirmed diagnosis of urological malignancy.
Proportion of potentially avoidable invasive procedures in AHG | At least 12 months from study inclusion.
  Percentage of invasive diagnostic procedures (e.g., cystoscopy, CT-urography) in the Acute Hemorrhagic Cystitis Group (AHG) that could have been avoided based on study findings.
Sensitivity and specificity of AHC classification | At least 12 months from study inclusion.
  Accuracy of the acute hemorrhagic cystitis (AHC) clinical classification in predicting urological malignancy, measured by sensitivity and specificity.

CONTACTS AND LOCATIONS:
Overall Officials: Suleiman Abuhasanein, Principal Investigator — Department of Urology, Institute of Clinical Science, Sahlgrenska Academy, University of Gothenburg
Locations (1):
- Uddevalla Hospital, Uddevalla, Sweden

IPD SHARING:
Plan to Share IPD: Undecided
At this time, no final decision has been made regarding sharing of individual participant data (IPD). Any future sharing would require appropriate ethical approvals, participant consent, and compliance with data protection regulations.